CLINICAL TRIAL: NCT02864953
Title: Randomized, Double-Blind, Placebo-Controlled, Parallel-Group, Multicenter, Phase 3 Study to Evaluate the Efficacy and Safety of Intravenous BIIB093 (Glibenclamide) for Severe Cerebral Edema Following Large Hemispheric Infarction
Brief Title: Phase 3 Study to Evaluate the Efficacy and Safety of Intravenous BIIB093 (Glibenclamide) for Severe Cerebral Edema Following Large Hemispheric Infarction
Acronym: CHARM
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Early completed to operational challenges and other strategic considerations, not for efficacy or safety reasons
Sponsor: Remedy Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 252LH301; RPI 301 (Other: Remedy Pharmaceuticals); 2017-004854-41 (EudraCT Number); NCT04950972 (obsolete NCT alias)
Record Dates: First submitted 2016-07-12; First posted 2016-08-12 (Estimated); Results first posted 2024-01-09 (Actual); Last update posted 2024-11-25 (Actual); Status verified 2024-11

CONDITIONS: Brain Edema; Stroke, Acute
Keywords: Infarction; Cerebrovascular Disorders; Brain Diseases; Pathological Processes Necrosis; Central Nervous System Diseases; Vascular Diseases; Cardiovascular Diseases; Glyburide; Hypoglycemic Agents; Physiological Effects of Drugs
MeSH Terms: conditions — Brain Edema; Stroke; Infarction; Cerebrovascular Disorders; Brain Diseases; Central Nervous System Diseases; Vascular Diseases; Cardiovascular Diseases | interventions — Glyburide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- BIIB093 (Experimental): BIIB093 administered as a bolus followed by continuous intravenous (IV) infusion over 72 hours.
  Interventions: Drug: BIIB093
- Placebo (Placebo Comparator): Placebo administered as a bolus followed by continuous intravenous (IV) infusion over 72 hours.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: BIIB093 — Administered as specified in the treatment arm.
  Other Names: glibenclamide; glibenclamide intravenous (IV); glyburide; CIRARA
  Arms: BIIB093
Drug: Placebo — Administered as specified in the treatment arm.
  Arms: Placebo

SUMMARY:
The primary objective of Part 1 of the study is to determine if BIIB093 improves functional outcome at Day 90 as measured by the modified Rankin Scale (mRS) when compared with placebo in participants with Large Hemispheric Infarction (LHI). The secondary objectives of Part 1 of the study are to determine if BIIB093 improves overall survival at Day 90 when compared with placebo, if BIIB093 improves functional outcome at Day 90 on the mRS dichotomized 0-4 vs. 5-6 when compared with placebo, if BIIB093 reduces midline shift at 72 hours (or at time of decompressive craniectomy [DC] or comfort measures only [CMO], if earlier) when compared with placebo, and to evaluate the safety and tolerability of BIIB093 in participants with LHI.

The objectives of Part 2 of the study are to evaluate long-term disability following LHI, to evaluate long-term outcome measures of clinical function, quality of life, and healthcare utilization, and to assess the safety of BIIB093 in subjects with LHI during the follow-up period.

ELIGIBILITY:
Inclusion Criteria:

1. A clinical diagnosis of acute ischemic stroke in the middle cerebral artery (MCA) territory.
2. A large hemispheric infarction defined as; lesion volume of 80 to 300 centimeters cubed (cm^3) on magnetic resonance imaging (MRI) diffusion-weighted imaging (DWI), or computed tomography perfusion (CTP), or an Alberta Stroke Program Early CT Score (ASPECTS) of 1 to 5 with involvement of at least 2 defined cortical regions.
3. Screening National Institutes of Health Stroke Scale (NIHSS) >=10.
4. At the time of randomization, and in the Investigator's judgement, it must be feasible for study drug treatment infusion to be initiated no later than 10 hours after time of symptom onset, if known, or the time last known normal.

   * Participants who wake with stroke may be included if neurological and other exclusion criteria are satisfied. The time of stroke onset is to be taken as the midpoint between sleep onset (or last known to be normal) and time of waking.
5. For participants who receive thrombectomy, inclusion into the study must be based on post-thrombectomy MRI-DWI.

Exclusion Criteria:

1. Participant is likely to have supportive care withdrawn on the first day.
2. Commitment to decompressive craniectomy (DC) prior to enrollment.
3. Evidence of concurrent infarction in the contralateral hemisphere sufficiently serious so as to affect functional outcome.

NOTE: Other protocol defined Inclusion/Exclusion criteria may apply

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 535 (Actual)
Dates: Start 2018-08-29 (Actual); Primary Completion 2023-08-18 (Actual); Study Completion 2023-08-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Remedy Pharmaceuticals
Locations (250):
- United States (74):
  - Barrow Neurological Institute, Phoenix, Arizona
  - Arizona Board of Regents, University of Arizona, Tucson, Arizona
  - Stanford Stroke Center, Palo Alto, California
  - University of California Davis Health System, Sacramento, California
  - UCSD Health-La Jolla, San Diego, California
  - University of Colorado Hospital, Aurora, Colorado
  - Yale New Haven Hospital, New Haven, Connecticut
  - University of Florida-Gainsville, Gainesville, Florida
  - Lyerly Neurosurgery Baptist Health, Jacksonville, Florida
  - University of Florida, Jacksonville, Jacksonville, Florida
  - University of South Florida, Tampa, Florida
  - Grady Memorial Hospital, Atlanta, Georgia
  - Augusta University, Augusta, Georgia
  - The Queens Medical Center, Honolulu, Hawaii
  - Rush University Medical Center, Chicago, Illinois
  - University of Kansas Medical Center Research Institute, Inc., Kansas City, Kansas
  - University of Louisville, Louisville, Kentucky
  - Ochsner Clinic Foundation, New Orleans, Louisiana
  - Maine Medical Center, Portland, Maine
  - University of Maryland, Baltimore, Maryland
  - Sinai Hospital of Baltimore, Baltimore, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts
  - Brigham and Woman's Hospital, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Inc., Jamaica Plain, Massachusetts
  - UMASS Memorial Medical Center, Worcester, Massachusetts
  - Henry Ford Hospital, Detroit, Michigan
  - St. John's Hospital, Detroit, Michigan
  - Fairview Southdale Hospital, Edina, Minnesota
  - Saint Luke's Hospital of Kansas City, Kansas City, Missouri
  - Saint Louis University, St Louis, Missouri
  - Washington University Physicians, St Louis, Missouri
  - JFK Medical Center, Edison, New Jersey
  - Jersey Shore University Medical Center, Neptune City, New Jersey
  - Rutgers - Robert Wood Johnson Medical School, New Brunswick, New Jersey
  - Valley Hospital, Ridgewood, New Jersey
  - University of New Mexico, Albuquerque, New Mexico
  - University of Buffalo, Buffalo, New York
  - Northwell Health, Manhasset, New York
  - NYU Langone Medical Center, New York, New York
  - Mount Sinai Hospital, New York, New York
  - Columbia University Hervert Irving Comprehensive Cancer Center, New York, New York
  - University of Rochester Medical Center, Rochester, New York
  - SUNY Upstate Medical Center, Syracuse, New York
  - UNC Hospitals, Chapel Hill, North Carolina
  - Atrium Health Carolinas Medical Center, Charlotte, North Carolina
  - Duke University Medical Center, Durham, North Carolina
  - Guilford Neurologic Research, PA, Greensboro, North Carolina
  - Novant Health Forsyth Medical Center, Winston-Salem, North Carolina
  - Wake Forest Baptist Health Sciences, Winston-Salem, North Carolina
  - Summa Health System, Akron, Ohio
  - University of Cincinnati, Cincinnati, Ohio
  - University Hospitals Cleveland Medical Center, Cleveland, Ohio
  - The Cleveland Clinic Foundation, Cleveland, Ohio
  - Ohio State Univ College Of Medicine, Columbus, Ohio
  - Miami Valley Hospital South, Dayton, Ohio
  - ProMedica Toledo Hospital, Toledo, Ohio
  - Ascension St. John, Tulsa, Oklahoma
  - Providence Brain and Spine Institute, Portland, Oregon
  - Oregon Health & Science University, Portland, Oregon
  - Lehigh Valley Hospital - Cedar Crest, Allentown, Pennsylvania
  - Penn State University Milton S. Hershey Medical Center, Hershey, Pennsylvania
  - University of Pennsylvania Health System, Philadelphia, Pennsylvania
  - Allegheny General Hospital, Pittsburgh, Pennsylvania
  - University of Pittsburgh School of Medicine, Pittsburgh, Pennsylvania
  - Rhode Island Hospital Warren Alpert Medical School Brown University, Providence, Rhode Island
  - Erlanger Health System, Chattanooga, Tennessee
  - University of Tennessee Health Sciences Center, Memphis, Tennessee
  - TriStar Skyline Medical Center, Nashville, Tennessee
  - Vanderbilt Medical Center, Nashville, Tennessee
  - St.David's HealthCare Office of Research, Austin, Texas
  - Valley Baptist Medical Center, Harlingen, Texas
  - University of Utah Neurology, Salt Lake City, Utah
  - University of Washington School of Medicine, Seattle, Washington
  - University Hospital and UW Health Clinics, Madison, Wisconsin
- Australia (9):
  - Liverpool Hospital, Liverpool, New South Wales
  - John Hunter Hospital, New Lambton Heights, New South Wales
  - Royal North Shore Hospital, St Leonards, New South Wales
  - Princess Alexandra Hospital, Woolloongabba, Queensland
  - Royal Adelaide Hospital, Adelaide, South Australia
  - Monash Medical Centre, Clayton, Victoria
  - The Alfred Hospital, Melbourne, Victoria
  - Royal Melbourne Hospital, Parkville, Victoria
  - Sunshine Hospital, St Albans, Victoria
- Belgium (4):
  - Universitair Ziekenhuis Gent, Ghent, East Flanders
  - UZ Leuven, Leuven, Flemish Brabant
  - CHU UCL Namur, Yvoir, Namur
  - Clinique CHC MontLégia, Liège
- Brazil (6):
  - HGF - Hospital Geral de Fortaleza, Fortaleza, Ceará
  - Hospital do Rocio, Campo Largo, Paraná
  - Hospital de Clínicas de Porto Alegre, Porto Alegre, Rio Grande do Sul
  - Clinica Neurológica e Neurocirúrgica de Joinville, Joinville, Santa Catarina
  - Hospital das Clínicas FMRP-USP, Ribeirão Preto, São Paulo
  - Hospital Sao Paulo, São Paulo, São Paulo
- Canada (2):
  - Foothills Medical Centre, Calgary, Alberta
  - University of Alberta Hospital, Edmonton, Alberta
- China (25):
  - Anhui Provincial Hospital, Hefei, Anhui
  - Xuanwu Hospital Capital Medical University, Beijing, Beijing Municipality
  - Beijing Tiantan Hospital, Capital Medical University, Beijing, Beijing Municipality
  - Peking University Third Hospital, Beijing, Beijing Municipality
  - Beijing Tiantan Hospital, Capital Medical University, Beijing, Bejing
  - The First Affiliated Hospital of Sun Yat-sen University, Guangzhou, Guangdong
  - The Second Affiliated Hospital of Guangzhou Medical University, Guangzhou, Guangdong
  - Hainan General Hospital, Haikou, Hainan
  - Tongji Hospital, Tongji Medical College, Huazhong University of Science & Technology, Wuhan, Hubei
  - Renmin Hospital, Wuhan University, Wuhan, Hubei
  - Huai'an First People's Hospital, Huai'an, Jiangsu
  - Zhongda Hospital Southeast University, Nanjing, Jiangsu
  - The Second Affiliated Hospital of Nanjing Medical University, Nanjing, Jiangsu
  - Affiliated Hospital of Nantong University, Nantong, Jiangsu
  - The Affiliated Hospital of Xuzhou Medical College, Xuzhou, Jiangsu
  - The Second Affiliated Hospital of Soochow University, Suzhou, Jiangsushe
  - Jiangxi Provincial People's Hospital, Nanchang, Jiangxi
  - The First Affiliated Hospital of Nanchang University, Nanchang, Jiangxi
  - Jiangxi Pingxiang People's Hospital, Pingxiang, Jiangxi
  - The First Hospital of Jilin University, Changchun, Jilin
  - Huashan Hospital, Fudan University, Shanghai, Shanghai Municipality
  - The Second Affiliated Hospital of Xi'an Jiaotong University（Xibei Hospital), Xi’an, Shanxi
  - Army Specialty Medical Center of The Chinese People's Liberation Army, Chongqing, Sichuan
  - Tianjin Medical University General Hospital, Tianjin, Tianjin Municipality
  - Sir Run Run Shaw Hospital, Zhejiang University School of Medicine, Hangzhou, Zhejiang
- Croatia (3):
  - General Hospital Varazdin, Varaždin, Croatia Proper
  - Clinical Hospital 'Sestre Milosrdnice', Zagreb, Croatia Proper
  - Clinical Hospital Centar Zagreb, Zagreb, Croatia Proper
- Czechia (6):
  - Fakultni nemocnice Ostrava, Ostrava, Moravian-Silesian
  - Fakultni nemocnice Brno, Brno, Moravia
  - Fakultni nemocnice u sv. Anny v Brne, Brno, Moravia
  - Fakultni nemocnice Kralovske Vinohrady, Prague, Prague
  - Fakultni nemocnice v Motole, Prague, Prague
  - Fakultni nemocnice Hradec Kralove, Hradec Králové
- Denmark (3):
  - Copenhagen University Hospital and Glostrup Hospital, Copenhagen, Copenhagen City
  - Bispebjerg og Frederiksberg Hospital, Copenhagen NV, Copenhagen City
  - Sjællands Universitetshospital, Roskilde, Østsjælland
- Finland (2):
  - Helsinki University Hospital, Helsinki, Southern
  - Turun yliopistollinen keskussairaala, Turku, Western
- France (9):
  - CHU CAEN - Hôpital de la Côte de Nacre, Caen, Calvados
  - CHU Besançon - Hôpital Jean Minjoz, Besançon, Doubs
  - CHU de Brest - Hôpital de la Cavale Blanche, Brest, Finistere
  - Groupe Hospitalier Pellegrin - Hôpital Pellegrin, Bordeaux, Gironde
  - CHU Rennes - Hopital Pontchaillou, Rennes, Ille-et-Vilaine
  - CHU Nantes - Hopital Nord Laënnec, Saint-Herblain, Loire Atlantique
  - CHU Nancy - Hôpital Central, Nancy, Meurthe Et Moselle
  - Hopital Roger Salengro - CHU Lille, Lille, Nord
  - Hôpital Bicêtre, Le Kremlin-Bicêtre, Val De Marne
- Germany (12):
  - Universitaetsklinikum Freiburg, Freiburg im Breisgau, Baden-Wurttemberg
  - Klinikum Augsburg, Augsburg, Bavaria
  - Rhon-Klnikum Campus Bad Neustadt, Bad Neustadt Saale, Bavaria
  - Universitaetsklinikum Erlangen, Erlangen, Bavaria
  - Klinikum der Johann Wolfgang Goethe-Universitaet, Frankfurt am Main, Hesse
  - Klinikum Frankfurt Hoechst GmbH, Frankfurt am Main, Hesse
  - Klinikum Kassel GmbH, Kassel, Hesse
  - Universitaetsklinikum Essen, Essen, North Rhine-Westphalia
  - Universitaetsklinikum Muenster, Münster, North Rhine-Westphalia
  - Klinikum Altenburger Land GmbH, Altenburg, Thuringia
  - Universitaetsklinikum Jena, Jena, Thuringia
  - Universitaetsklinikum Carl Gustav Carus TU Dresden, Dresden
- Hungary (6):
  - Pest Megyei Flor Ferenc Korhaz, Kistarcsa, Budapest
  - Szegedi Tudomanyegyetem Szent-Gyorgyi Albert Klinikai Kozpont, Szeged, Csongrád-Csanád
  - Petz Aladar Egyetemi Oktato Korhaz, Győr, Győr-Moson-Sopron
  - Somogy Megyei Kaposi Mor Oktato Korhaz, Kaposvár, Somogy County
  - SzSzB Megyei Korhazak es Egyetemi Oktatokorhaz, Nyíregyháza, Szabolcs-Szatmár-Bereg
  - Semmelweis Egyetem, Budapest
- Israel (6):
  - Rabin MC, Petah Tikva, Central District
  - Soroka University Medical Center, Beersheba, Southern District
  - Rambam Health Care Center, Haifa
  - Shaare Zedek, Jerusalem
  - Hadassah University Hospital - Ein Kerem, Jerusalem
  - Tel Aviv Sourasky Medical Center, Tel Aviv
- Italy (11):
  - Istituto Clinico Humanitas, Rozzano, Milano
  - Azienda Ospedaliera Universitaria Policlinico Tor Vergata, Rome, Roma
  - Policlinico Umberto I, Rome, Roma
  - Azienda Ospedaliera Sant'Andrea-Università di Roma La Sapienza, Rome, Roma
  - Azienda Socio Sanitaria Territoriale degli Spedali Civili di Brescia (Presidio Spedali Civili), Brescia
  - Azienda Ospedaliera Universitaria Careggi, Florence
  - IRCCS Ospedale Policlinico San Martino, Genova
  - Fondazione IRCCS CA' Granda Ospedale Maggiore Policlinico, Milan
  - Ospedale San Raffaele, Milan
  - Azienda Socio Sanitaria Territoriale Niguarda (Grande Ospedale Metropolitano Niguarda), Milan
  - A.O.U. Senese Policlinico Santa Maria alle Scotte, Siena
- Japan (28):
  - Toyota Memorial Hospital, Toyota-shi, Aichi-ken
  - Hachinohe Red Cross Hospital, Hachinohe-shi, Aomori
  - Kimitsu Chuo Hospital, Kisarazu-shi, Chiba
  - NHO Kyushu Medical Center, Fukuoka, Fukuoka
  - Chiyukai Fukuoka Wajiro Hospital, Fukuoka, Fukuoka
  - Chiyukai Fukuoka Shinmizumaki Hospital, Onga-gun, Fukuoka
  - Chiyukai Shin Yukuhashi Hospital, Yukuhashi-shi, Fukuoka
  - Southern Tohoku General Hospital, Koriyama-shi, Fukushima
  - Gifu Prefectural General Medical Center, Gifu, Gifu
  - Showakai Brain Attack Center Ota Memorial Hospital, Fukuyama-shi, Hiroshima
  - Asahikawa Red Cross Hospital, Asahikawa-shi, Hokkaido
  - Ohnishi Neurological Center, Akashi-shi, Hyōgo
  - Kobe City Hospital Organization Kobe City Medical Center General Hospital, Kobe, Hyōgo
  - Tsuchiura Kyodo General Hospital, Tsuchiura-shi, Ibaraki
  - Iwate Prefectural Central Hospital, Morioka, Iwate
  - St. Marianna University Hospital, Kawasaki-shi, Kanagawa
  - NHO Sendai Medical Center, Sendai, Miyagi
  - Kurashiki Central Hospital, Kurashiki-shi, Okayama-ken
  - Okayama City General Medical Center Okayama City Hospital, Okayama, Okayama-ken
  - Rinku General Medical Center, Izumisano, Osaka
  - National Cerebral and Cardiovascular Center, Suita, Osaka
  - Saitama Medical University International Medical Center, Hidaka-shi, Saitama
  - Nippon Medical School Hospital, Bunkyō City, Tokyo-To
  - Tokyo Metropolitan Tama Medical Center, Fuchu-shi, Tokyo-To
  - Kyorin University Hospital, Mitaka-shi, Tokyo-To
  - NHO Minami Wakayama Medical Center, Tanabe-shi, Wakayama
  - Yamaguchi University Hospital, Ube-shi, Yamaguchi
  - Yamanashi Prefectural Central Hospital, Kofu, Yamanashi
- Lithuania (3):
  - Hospital of Lithuanian University of Health Sciences Kaunas Clinics, Kaunas
  - Republican Vilnius University Hospital, Public Institution, Vilnius
  - Vilnius University Hospital Santariskiu Clinic, Public Institution, Vilnius
- Portugal (7):
  - Centro Hospitalar de Entre o Douro e Vouga, E.P.E. - Hospital de São Sebastião, Santa Maria da Feira, Aveiro District
  - Unidade Local de Saúde de Matosinhos, E.P.E. - Hospital Pedro Hispano, Matosinhos Municipality, Porto District
  - Hospital Garcia de Orta, EPE, Almada, Setúbal District
  - Centro Hospitalar e Universitário de Coimbra E.P.E. - Hospitais da Universidade de Coimbra, Coimbra
  - Centro Hospitalar de Lisboa Ocidental, E.P.E. - Hospital de Egas Moniz, Lisbon
  - Centro Hospitalar de Lisboa Norte, E.P.E. - Hospital de Santa Maria, Lisbon
  - Centro Hospitalar de São João, E.P.E, Porto
- Russia (5):
  - SBEI HPE 'Kazan State Medical University' of the MoH of the RF, Kazan', Respublka Tatarstan
  - Saint-Petersburg Scientific-Research Institute of Emergency Care, Saint Petersburg, Sankt-Peterburg
  - SPb SBIH 'City Hospital # 26', Saint Petersburg, Sankt-Peterburg
  - SHI "Territorial Clinical Hospital #1 n.a. S.V. Ochapovsky", Krasnodar
  - SBIH of Moscow 'City Clinical Hospital # 1 n. a. N. I. Pirogov', Moscow
- South Korea (4):
  - Seoul National University Bundang Hospital, Seongnam-si, Gyeonggi-do
  - Kyungpook National University Hospital, Daegu, Gyeongsangnam-do
  - Dong-A University Hospital, Busan
  - Asan Medical Center, Seoul
- Spain (12):
  - Hospital Universitari de Bellvitge, L'Hospitalet de Llobregat, Barcelona
  - Hospital Universitario Reina Sofia, Córdoba, Córdoba
  - Complejo Hospitalario Universitario de Santiago, Santiago de Compostela, La Coruña
  - Hospital Regional Universitario de Malaga, Málaga, Málaga
  - Hospital del Mar, Barcelona
  - Hospital Universitari Vall d'Hebron, Barcelona
  - Hospital Universitari de Girona Dr Josep Trueta, Girona
  - Hospital Universitario Ramon y Cajal, Madrid
  - Hospital Universitario Virgen del Rocio, Seville
  - Hospital Universitario Virgen Macarena, Seville
  - Hospital Universitari i Politecnic La Fe, Valencia
  - Hospital Clinico Universitario de Valladolid, Valladolid
- Switzerland (2):
  - Ospedale Regionale di Lugano, Lugano, Canton Ticino
  - Inselspital - Universitaetsspital Bern, Bern
- Taiwan (4):
  - Kaohsiung Chang Gung Memorial Hospital, Kaohsiung City
  - National Cheng Kung University Hospital, Tainan
  - National Taiwan University Hospital, Taipei
  - Chang Gung Memorial Hospital,Linkou, Taoyuan District
- United Kingdom (7):
  - Addenbrooke's Hospital, Cambridge, Cambridgeshire
  - King's College Hospital, London, Greater London
  - Imp Coll Health Nhst 1, London, Greater London
  - The National Hospital for Neurology & Neurosurgery, London, Greater London
  - Nottingham University Hospitals City Campus, Nottingham, Nottinghamshire
  - Queen Elizabeth University Hospital Campus, Glasgow, Strathclyde
  - Newcastle University- Clinical Ageing Research Unit, Newcastle upon Tyne, Tyne & Wear

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Sheth KN, Albers GW, Saver JL, Campbell BCV, Molyneaux BJ, Hinson HE, Cordonnier C, Steiner T, Toyoda K, Wintermark M, Littauer R, Collins J, Lucas N, Nogueira RG, Simard JM, Wald M, Dawson K, Kimberly WT; CHARM Trial investigators. Intravenous glibenclamide for cerebral oedema after large hemispheric stroke (CHARM): a phase 3, double-blind, placebo-controlled, randomised trial. Lancet Neurol. 2024 Dec;23(12):1205-1213. doi: 10.1016/S1474-4422(24)00425-3. PMID 39577921
- [Derived] Shu L, Zhang W, Yaghi S, Grilli A, de Havenon A, Barrett KM, Johnston KC, Goldstein ED. Prestroke and Poststroke Sulfonylurea Exposure and Functional Outcomes: A Post Hoc Analysis of the SHINE Trial. Stroke. 2023 Sep;54(9):e415-e416. doi: 10.1161/STROKEAHA.123.043496. Epub 2023 Jul 14. No abstract available. PMID 37449423

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled at investigative sites in the United States, Brazil, China, Spain, Japan, Australia, Portugal, Germany, United Kingdom, Finland, Canada, Israel, France, Taiwan, Hungary, Czech Republic, Italy, Belgium, Lithuania, Russia and South Korea from 29 August 2018 to 18 August 2023.
Pre-assignment Details: A total of 535 participants were enrolled and randomised, out of which 518 participants were dosed with BIIB093 or a matching placebo.
Groups:
- Placebo: Participants were administered with BIIB093 matching placebo as an intravenous (IV) bolus on Day 1 followed by a continuous IV infusion for over 72 hours.
- BIIB093: Participants were administered with BIIB093 as an IV bolus on Day 1 followed by continuous IV infusion for over 72 hours.
Period: Overall Study
Arm/Group | Placebo | BIIB093
Started | 268 | 267
Completed | 215 | 213
Not Completed | 53 | 54
Not completed — Adverse Event | 22 | 19
Not completed — Withdrawal by Subject | 1 | 0
Not completed — Physician Decision | 4 | 2
Not completed — Death | 3 | 13
Not completed — Reason not specified | 14 | 12
Not completed — Withdrew Prior to Dosing | 9 | 8

BASELINE CHARACTERISTICS:
Population: The Intent-to-treat (ITT) population included all randomized participants.
Groups:
- Placebo: Participants were administered with BIIB093 matching placebo as an IV bolus on Day 1 followed by a continuous IV infusion for over 72 hours.
- Total: Total of all reporting groups
Arm/Group | Placebo | BIIB093 | Total
Number analyzed (Participants) | 268 | 267 | 535
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.6 (10.81) | 60.5 (11.17) | 61.1 (11)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 104 | 98 | 202
  Male | 164 | 169 | 333
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Ethnicity: Missing | 1 | 2 | 3
  Ethnicity: Hispanic or Latino | 36 | 41 | 77
  Ethnicity: Not Hispanic or Latino | 228 | 223 | 451
  Ethnicity: Not reported | 3 | 1 | 4
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: Missing | 3 | 2 | 5
  Race: American Indian or Alaska Native | 1 | 1 | 2
  Race: Asian | 53 | 51 | 104
  Race: Black or African American | 21 | 19 | 40
  Race: Native Hawaiian or Other Pacific Islander | 2 | 0 | 2
  Race: White | 173 | 177 | 350
  Race: Not reported due to confidentiality regulations | 3 | 1 | 4
  Race: Other | 12 | 16 | 28

OUTCOME MEASURES:

1. Primary Outcome: Part 1: Percentage of Participants With Improvement in Functional Outcome at Day 90 Assessed Via the Modified Rankin Scale (mRS)
Description: The mRS measures the degree of functional independence following stroke. In this study, 7-category ordinal mRS scale was condensed to the following 5-categories: 0/1, 2, 3, 4, 5/6 where 0 and 1 reflect no disability and near-normal functioning while 5 and 6 represent severe disability and death, respectively.
Time Frame: Day 90
Population: The modified intent to treat (mITT) population included participants aged 18 to 70 years (inclusive) at the time of randomization, who had received any study drug, and who had at least 1 post-baseline mRS before or at Day 90 visit. Here, 'Overall number of participants analyzed' signifies the number of participants with data available for outcome measure analysis.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | BIIB093
Number analyzed (Participants) | 214 | 217
percentage of participants
  Score: 0/1 | 1.4 | 3.2
  Score: 2 | 2.8 | 5.1
  Score: 3 | 12.6 | 12.0
  Score: 4 | 25.2 | 23.5
  Score: 5/6 | 57.9 | 56.2
Statistical Analysis 1: Comparison: Placebo vs BIIB093; Test type: Superiority; p = 0.4150, Regression, Logistic — P-value was analyzed by ordinal logistic regression adjusting for covariates: region, and IRT stratification factors including rtPA usage (yes/no), thrombectomy usage (yes/no), use of ASPECTS for screening (yes/no), baseline NIHSS (<=20 vs. >20); Odds Ratio (OR) = 1.17, 95% CI 2-sided [0.80 to 1.71]

2. Secondary Outcome: Part 1: Time to All-Cause Death Through Day 90
Description: Time to all-cause death is defined as the time from randomization to the time of death.
Time Frame: Randomization up to Day 90
Population: The mITT population included participants aged 18 to 70 years (inclusive) at the time of randomization, who received any study drug, and who had at least 1 post-baseline mRS before or at the Day 90 visit. Here, 'Overall number of participants analyzed' signifies number of participants with data available for outcome measure analysis.
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Placebo | BIIB093
Number analyzed (Participants) | 214 | 217
days | NA [37 to NA] — Median and upper limit of inter quartile range were not reached due to insufficient number of participants with events. | NA [18 to NA] — Median and upper limit of inter quartile range were not reached due to insufficient number of participants with events.

3. Secondary Outcome: Part 1: Percentage of Participants Who Achieved mRS 0-4 at Day 90
Description: The mRS measures the degree of functional independence following stroke. In this study, the 7-category ordinal mRS scale was condensed to the following 5-categories: 0/1, 2, 3, 4, 5/6 where 0 and 1 reflect no disability and near-normal functioning while 5 and 6 represent severe disability and death, respectively.
Time Frame: Day 90
Population: as for outcome 2
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | BIIB093
Number analyzed (Participants) | 214 | 217
percentage of participants | 41.6 | 42.9
Statistical Analysis 1: Comparison: Placebo vs BIIB093; Test type: Superiority; p = 0.7413, Regression, Logistic — A logistic regression model was used to estimate an odds ratio (and 95% CI) of improvement on the mRS dichotomized as 0-4 vs. 5-6 at Day 90; Odds Ratio (OR) = 1.07, 95% CI 2-sided [0.72 to 1.60]

4. Secondary Outcome: Part 1: Midline Shift at 72 Hours as Assessed by Non-contrast Computed Tomography (NCCT) or Magnetic Resonance Imaging (MRI)
Description: Midline shift is the perpendicular distance between the septum pellucidum and the line drawn between the anterior and posterior attachments of the falx to the inner table of the skull.
Time Frame: At 72 hours
Population: The mITT population included participants aged 18 to 70 years (inclusive) at the time of randomization, who received any study drug, and who had at least 1 post-baseline mRS before or at the Day 90 visit. Here, 'Overall number of participants analyzed' signifies the number of participants with data available for outcome measure analysis.
Measure: Mean (Standard Deviation); unit: millimeters (mm)
Arm/Group | Placebo | BIIB093
Number analyzed (Participants) | 150 | 155
millimeters (mm) | 6.32 (4.760) | 7.02 (4.565)
Statistical Analysis 1: Comparison: Placebo vs BIIB093; Test type: Superiority; p = 0.1242, ANOVA — Analysis of Variance (ANOVA) was used to compare the two study arms to assess the treatment effects on midline shift; Mean Difference (Final Values) = 0.82, 95% CI 2-sided [-0.23 to 1.87]

5. Secondary Outcome: Part 1: Percentage of Participants With Adverse Events (AEs) and Serious Adverse Events (SAEs)
Description: An AE is any untoward medical occurrence in a participant or clinical investigation participant administered a pharmaceutical product and that does not necessarily have a causal relationship with this treatment. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with the use of a medicinal (investigational) product, whether or not related to the medicinal (investigational) product. A SAE is any untoward medical occurrence that at any dose results in death, life-threatening event, requires inpatient hospitalization, significant disability/incapacity or congenital anomaly.
Time Frame: From the signing of informed consent up to the last follow-up visit (up to 4 years 11 months)
Population: The safety population included all participants who were enrolled and had received any portion of the infusion of study treatment (placebo or BIIB093). Here, 'Overall number of participants analyzed' signifies the number of participants with data available for outcome measure analysis.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | BIIB093
Number analyzed (Participants) | 259 | 259
percentage of participants
  AEs | 95.4 | 97.3
  SAEs | 68.3 | 76.8

ADVERSE EVENTS:
Time Frame: From the signing of informed consent up to the last follow-up visit (up to 4 years 11 months)
Description: The safety population included all participants who were enrolled and had received any portion of the infusion of study treatment (placebo or BIIB093).
Groups:
- Placebo: Participants were administered with BIIB093 matching placebo as an IV bolus followed by a continuous IV infusion for over 72 hours.
- BIIB093: Participants were administered with BIIB093 as an IV bolus followed by continuous IV infusion for over 72 hours.
Arm/Group | Placebo | BIIB093
All-Cause Mortality (participants affected / at risk) | 97/259 | 103/259
Serious Adverse Events (participants affected / at risk) | 177/259 | 199/259
Other Adverse Events (participants affected / at risk) | 199/259 | 201/259
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=259) | BIIB093 (N=259)
Anaemia (Blood and lymphatic system disorders) | 3 | 2
Blood loss anaemia (Blood and lymphatic system disorders) | 1 | 0
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 0 | 1
Neutropenia (Blood and lymphatic system disorders) | 1 | 0
Acute coronary syndrome (Cardiac disorders) | 1 | 0
Acute myocardial infarction (Cardiac disorders) | 2 | 1
Atrial fibrillation (Cardiac disorders) | 4 | 2
Atrial flutter (Cardiac disorders) | 1 | 0
Bradycardia (Cardiac disorders) | 1 | 1
Cardiac arrest (Cardiac disorders) | 5 | 5
Cardiac failure (Cardiac disorders) | 2 | 1
Cardiac failure congestive (Cardiac disorders) | 2 | 0
Cardiac ventricular thrombosis (Cardiac disorders) | 0 | 2
Cardio-respiratory arrest (Cardiac disorders) | 2 | 1
Cardiogenic shock (Cardiac disorders) | 1 | 1
Cardiomyopathy (Cardiac disorders) | 1 | 0
Cardiopulmonary failure (Cardiac disorders) | 1 | 2
Dilated cardiomyopathy (Cardiac disorders) | 1 | 0
Myocardial infarction (Cardiac disorders) | 1 | 1
Myocardial ischaemia (Cardiac disorders) | 1 | 0
Pericardial effusion (Cardiac disorders) | 1 | 0
Sinus tachycardia (Cardiac disorders) | 0 | 1
Tachycardia paroxysmal (Cardiac disorders) | 0 | 1
Ventricular fibrillation (Cardiac disorders) | 1 | 1
Ventricular tachycardia (Cardiac disorders) | 2 | 0
Atrial septal defect (Congenital, familial and genetic disorders) | 1 | 0
Diabetes insipidus (Endocrine disorders) | 1 | 1
Inappropriate antidiuretic hormone secretion (Endocrine disorders) | 0 | 1
Ascites (Gastrointestinal disorders) | 0 | 1
Colitis ulcerative (Gastrointestinal disorders) | 1 | 0
Constipation (Gastrointestinal disorders) | 0 | 1
Dysphagia (Gastrointestinal disorders) | 1 | 2
Gastritis (Gastrointestinal disorders) | 0 | 1
Ileus (Gastrointestinal disorders) | 1 | 1
Pelvic floor hernia (Gastrointestinal disorders) | 0 | 1
Retroperitoneal haematoma (Gastrointestinal disorders) | 0 | 1
Cardiac death (General disorders) | 1 | 0
Chest pain (General disorders) | 2 | 1
Death (General disorders) | 2 | 3
Malaise (General disorders) | 0 | 1
Multiple organ dysfunction syndrome (General disorders) | 1 | 1
Pyrexia (General disorders) | 0 | 3
Bile duct stone (Hepatobiliary disorders) | 1 | 0
Abdominal wall abscess (Infections and infestations) | 0 | 1
Acinetobacter infection (Infections and infestations) | 1 | 0
Bacterial infection (Infections and infestations) | 1 | 0
Bacterial sepsis (Infections and infestations) | 0 | 1
Cellulitis (Infections and infestations) | 0 | 1
Clostridium difficile colitis (Infections and infestations) | 0 | 3
Covid-19 (Infections and infestations) | 1 | 1
Covid-19 pneumonia (Infections and infestations) | 1 | 0
Cystitis (Infections and infestations) | 0 | 1
Cytomegalovirus enteritis (Infections and infestations) | 0 | 1
Device related infection (Infections and infestations) | 0 | 1
Enterobacter pneumonia (Infections and infestations) | 0 | 1
Enterococcal sepsis (Infections and infestations) | 1 | 0
Escherichia sepsis (Infections and infestations) | 1 | 2
Gas gangrene (Infections and infestations) | 0 | 1
Haematological infection (Infections and infestations) | 1 | 1
Klebsiella sepsis (Infections and infestations) | 1 | 0
Klebsiella urinary tract infection (Infections and infestations) | 1 | 0
Neurosyphilis (Infections and infestations) | 1 | 0
Pneumonia (Infections and infestations) | 18 | 13
Pneumonia aspiration (Infections and infestations) | 5 | 5
Pneumonia bacterial (Infections and infestations) | 1 | 5
Pneumonia haemophilus (Infections and infestations) | 1 | 1
Pneumonia klebsiella (Infections and infestations) | 1 | 0
Pneumonia staphylococcal (Infections and infestations) | 1 | 3
Post procedural infection (Infections and infestations) | 1 | 0
Postoperative wound infection (Infections and infestations) | 1 | 0
Proteus infection (Infections and infestations) | 1 | 1
Pseudomonal sepsis (Infections and infestations) | 1 | 0
Pulmonary sepsis (Infections and infestations) | 4 | 0
Pyelonephritis (Infections and infestations) | 0 | 1
Respiratory tract infection (Infections and infestations) | 0 | 1
Sepsis (Infections and infestations) | 4 | 6
Septic shock (Infections and infestations) | 4 | 6
Staphylococcal bacteraemia (Infections and infestations) | 2 | 1
Streptococcal abscess (Infections and infestations) | 1 | 0
Streptococcal sepsis (Infections and infestations) | 0 | 1
Tracheobronchitis (Infections and infestations) | 0 | 3
Urinary tract infection (Infections and infestations) | 4 | 6
Urinary tract infection pseudomonal (Infections and infestations) | 0 | 1
Urosepsis (Infections and infestations) | 1 | 4
Wound infection staphylococcal (Infections and infestations) | 2 | 0
Anastomotic ulcer haemorrhage (Injury, poisoning and procedural complications) | 0 | 1
Brain herniation (Injury, poisoning and procedural complications) | 16 | 19
Fall (Injury, poisoning and procedural complications) | 1 | 4
Hip fracture (Injury, poisoning and procedural complications) | 0 | 1
Intentional overdose (Injury, poisoning and procedural complications) | 1 | 1
Neurological procedural complication (Injury, poisoning and procedural complications) | 12 | 11
Post procedural haematoma (Injury, poisoning and procedural complications) | 0 | 2
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 0 | 2
Subdural haemorrhage (Injury, poisoning and procedural complications) | 0 | 1
Toxicity to various agents (Injury, poisoning and procedural complications) | 1 | 0
Anticoagulation drug level below therapeutic (Investigations) | 0 | 1
Neurological examination abnormal (Investigations) | 1 | 0
Cachexia (Metabolism and nutrition disorders) | 0 | 1
Decreased appetite (Metabolism and nutrition disorders) | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 1 | 0
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 1 | 1
Failure to thrive (Metabolism and nutrition disorders) | 1 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 1
Hypernatraemia (Metabolism and nutrition disorders) | 1 | 1
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 | 1
Hypoglycaemia (Metabolism and nutrition disorders) | 4 | 15
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 1
Metabolic acidosis (Metabolism and nutrition disorders) | 0 | 1
Gouty arthritis (Musculoskeletal and connective tissue disorders) | 0 | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Adenocarcinoma of colon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Cardiac myxoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Lung cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Ovarian clear cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Ovarian epithelial cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Pancreatic carcinoma metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Prostate cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Brain compression (Nervous system disorders) | 0 | 1
Brain oedema (Nervous system disorders) | 79 | 72
Brain stem haemorrhage (Nervous system disorders) | 0 | 1
Cerebellar haemorrhage (Nervous system disorders) | 0 | 1
Cerebral artery occlusion (Nervous system disorders) | 0 | 1
Cerebral haemorrhage (Nervous system disorders) | 1 | 1
Cerebral infarction (Nervous system disorders) | 8 | 10
Cerebral mass effect (Nervous system disorders) | 2 | 4
Cerebrovascular accident (Nervous system disorders) | 5 | 17
Cerebrovascular insufficiency (Nervous system disorders) | 0 | 1
Embolic cerebral infarction (Nervous system disorders) | 1 | 0
Epilepsy (Nervous system disorders) | 2 | 2
Facial paralysis (Nervous system disorders) | 1 | 0
Haemorrhage intracranial (Nervous system disorders) | 1 | 1
Haemorrhagic cerebellar infarction (Nervous system disorders) | 1 | 0
Haemorrhagic cerebral infarction (Nervous system disorders) | 2 | 1
Haemorrhagic transformation stroke (Nervous system disorders) | 16 | 14
Hydrocephalus (Nervous system disorders) | 1 | 0
Intensive care unit acquired weakness (Nervous system disorders) | 0 | 1
Ischaemic stroke (Nervous system disorders) | 3 | 8
Lacunar infarction (Nervous system disorders) | 1 | 0
Lacunar stroke (Nervous system disorders) | 1 | 0
Malignant middle cerebral artery syndrome (Nervous system disorders) | 1 | 2
Migraine (Nervous system disorders) | 0 | 1
Neurological decompensation (Nervous system disorders) | 0 | 3
Post stroke epilepsy (Nervous system disorders) | 0 | 4
Psychogenic seizure (Nervous system disorders) | 0 | 1
Seizure (Nervous system disorders) | 10 | 6
Status epilepticus (Nervous system disorders) | 4 | 1
Stroke in evolution (Nervous system disorders) | 6 | 14
Subarachnoid haemorrhage (Nervous system disorders) | 1 | 0
Subdural hygroma (Nervous system disorders) | 1 | 0
Device dislocation (Product Issues) | 0 | 1
Agitation (Psychiatric disorders) | 1 | 0
Confusional state (Psychiatric disorders) | 1 | 0
Delirium (Psychiatric disorders) | 1 | 0
Delirium tremens (Psychiatric disorders) | 0 | 1
Depression (Psychiatric disorders) | 0 | 1
Depression suicidal (Psychiatric disorders) | 0 | 2
Mental status changes (Psychiatric disorders) | 2 | 1
Suicide attempt (Psychiatric disorders) | 1 | 1
Acute kidney injury (Renal and urinary disorders) | 3 | 7
Renal failure (Renal and urinary disorders) | 2 | 0
Renal tubular necrosis (Renal and urinary disorders) | 0 | 1
Tubulointerstitial nephritis (Renal and urinary disorders) | 1 | 0
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 6 | 6
Aspiration (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Choking (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Chronic respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Laryngeal oedema (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Obstructive airways disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pneumomediastinum (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 8 | 8
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Respiratory acidosis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Respiratory arrest (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Respiratory depression (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 11 | 10
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 0 | 2
Arteriosclerosis (Vascular disorders) | 0 | 1
Circulatory collapse (Vascular disorders) | 1 | 1
Deep vein thrombosis (Vascular disorders) | 2 | 5
Haemodynamic instability (Vascular disorders) | 0 | 1
Hypertensive urgency (Vascular disorders) | 1 | 0
Hypotension (Vascular disorders) | 2 | 0
Peripheral artery occlusion (Vascular disorders) | 1 | 0
Peripheral artery thrombosis (Vascular disorders) | 1 | 0
Reperfusion injury (Vascular disorders) | 0 | 1
Shock (Vascular disorders) | 3 | 1
Thrombosis (Vascular disorders) | 0 | 1
Venous thrombosis (Vascular disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=259) | BIIB093 (N=259)
Anaemia (Blood and lymphatic system disorders) | 28 | 25
Leukocytosis (Blood and lymphatic system disorders) | 21 | 16
Atrial fibrillation (Cardiac disorders) | 22 | 17
Bradycardia (Cardiac disorders) | 13 | 13
Constipation (Gastrointestinal disorders) | 54 | 40
Diarrhoea (Gastrointestinal disorders) | 24 | 13
Dysphagia (Gastrointestinal disorders) | 6 | 13
Nausea (Gastrointestinal disorders) | 17 | 13
Vomiting (Gastrointestinal disorders) | 26 | 22
Pain (General disorders) | 8 | 14
Pyrexia (General disorders) | 57 | 66
Pneumonia (Infections and infestations) | 40 | 32
Pneumonia aspiration (Infections and infestations) | 14 | 15
Urinary tract infection (Infections and infestations) | 41 | 29
Electrocardiogram qt prolonged (Investigations) | 13 | 6
Hyperglycaemia (Metabolism and nutrition disorders) | 15 | 14
Hypernatraemia (Metabolism and nutrition disorders) | 23 | 26
Hypocalcaemia (Metabolism and nutrition disorders) | 11 | 13
Hypoglycaemia (Metabolism and nutrition disorders) | 8 | 31
Hypokalaemia (Metabolism and nutrition disorders) | 32 | 35
Hyponatraemia (Metabolism and nutrition disorders) | 18 | 18
Hypophosphataemia (Metabolism and nutrition disorders) | 23 | 14
Brain oedema (Nervous system disorders) | 28 | 28
Haemorrhagic transformation stroke (Nervous system disorders) | 24 | 16
Headache (Nervous system disorders) | 27 | 22
Acute kidney injury (Renal and urinary disorders) | 11 | 17
Urinary retention (Renal and urinary disorders) | 20 | 10
Deep vein thrombosis (Vascular disorders) | 9 | 16
Hypertension (Vascular disorders) | 13 | 7
Hypotension (Vascular disorders) | 18 | 14

LIMITATIONS AND CAVEATS:
Early termination of trial due to operational challenges and other strategic considerations, not for efficacy or safety reasons.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Our agreement is subject to confidentiality but generally the PI can publish, for noncommercial purposes only, results and methods of the trial, but no other Sponsor Confidential Information. PI must give Sponsor no less than 60 days to review any manuscript for a proposed publication and must delay publication for up to an additional 90 days thereafter if Sponsor needs to file any patent application to protect any of Sponsor's intellectual property contained in the proposed publication.

DOCUMENTS (2):
  • Study Protocol (2021-06-11): https://cdn.clinicaltrials.gov/large-docs/53/NCT02864953/Prot_000.pdf
  • Statistical Analysis Plan (2023-07-11): https://cdn.clinicaltrials.gov/large-docs/53/NCT02864953/SAP_001.pdf